CLINICAL TRIAL: NCT02764775
Title: Measuring Head Control Changes With 2d Video Analysis After Utilization of the Headpod in Children With Cerebral Palsy and Poor Head Control
Brief Title: Measuring Head Control Change With 2D Video Analysis After Utilization of Headpod in Children With Poor Head Control
Acronym: headpod
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Responsible Party: Principal Investigator, Julie Brown, PT, DPT, PCS, Texas Woman's University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17641
Record Dates: First submitted 2016-05-02; First posted 2016-05-06 (Estimated); Results first posted 2019-01-29 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: To Determine Efficacy of the Headpod; Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Quasi-experimental, one-way repeated measures design
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Headed utilization (Experimental): Use of Headpod for 6 months duration; 3 x per day for a minimum of 15 minutes each time;
  Interventions: Device: Headpod

INTERVENTIONS:
Device: Headpod — Adaptive equipment to assist with active head movements

SUMMARY:
Inclusion Criteria: children ages 2 to 14 years with poor head control and non progressive diagnoses. Exclusion criteria: significant change of status i.e. prolonged hospitalization, surgery; inability to tolerate using Headpod. Requires use of Headpod 3x per day for minimum of 15 minutes each time over a 6 month period. Log must be kept documenting usage of the Headpod. Video will be taken to document changes.

DETAILED DESCRIPTION:
Requires usage of the Headpod 3x per day for a minimum of 15 minutes each time. Usage required for 6 month period. Log must be kept documenting usage of the Headpod. Video will be taken on initial trial use, 1 week post trial use, at 3 months post utilization of the Headpod and at 6 months post utilization of the Headpod.

ELIGIBILITY:
Inclusion Criteria:

* non progressive diagnoses with poor head control

Exclusion Criteria:

* recent prolonged hospitalization; surgery, inability to tolerate wearing the Headpod

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie E Brown, DPT, Principal Investigator — Texas Woman's University
Locations (1):
- TWU School of Physical Therapy, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Headpod Utilization: Use of Headpod for 6 months duration; 3 x per day for a minimum of 15 minutes each time. Three measurements were taken: Prior to Headpod use, after 3 months of Headpod use and, after 6 months of Headpod use.
  Headpod: Adaptive equipment to assist with active head movements
Period: Overall Study
Arm/Group | Headpod Utilization
Started | 14 (All 14 participants were assigned to the Headpod utilization group.)
Completed | 8
Not Completed | 6
Not completed — Death | 1
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Groups:
- Headpod Utilization: Use of Headpod for 6 months duration; 3 x per day for a minimum of 15 minutes each time;
  Headpod: Adaptive equipment to assist with active head movements
Arm/Group | Headpod Utilization
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 7 [3 to 11]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14
Active head time [Mean (Standard Deviation); unit: seconds] — Amount of time in seconds the child was able to hold the head upright against gravity.
  seconds | 190.33 (42.31)

OUTCOME MEASURES:

1. Primary Outcome: Change in Head Holding Active Time From Baseline to 6 Months
Description: Active time in seconds holding head upright
Time Frame: baseline to 6 months
Population: Children ages 3 to 11 years
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Headpod Utilization
Number analyzed (Participants) | 14
Seconds | 83.63 (38.07)

ADVERSE EVENTS:
Time Frame: 1 year, 6 months
Description: All cause mortality: One child unexpectedly died 2 months into the study. The death was unrelated to Headpod use.
Arm/Group | Headed Utilization
All-Cause Mortality (participants affected / at risk) | 1/14
Serious Adverse Events (participants affected / at risk) | 1/14
Other Adverse Events (participants affected / at risk) | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Headed Utilization (N=14)
Death unrelated to participation in study (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No